CLINICAL TRIAL: NCT06683170
Title: Validity and Feasibility of the Pregnancy Monitoring Belt - a Clinical Pilot Study
Status: Not yet recruiting | Type: Observational
Sponsor: Anna Axelin (Other)
Responsible Party: Sponsor-Investigator, Anna Axelin, Professor, University of Turku
Organization: University of Turku (Other)
Other Study IDs: VARHA/12935/13.02.02/2024
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Validation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant women: Pregnant women wearing the pregnancy monitoring belt for two hours. In addition, the hospital patient monitor will be used to measure mother ECG, heart rate, breathing rate, oxygen saturation, blood pressure, contractions and fetal heart rate and movements.
- Healthcare professionals: Healthcare professionals participating in the pregnancy care.

SUMMARY:
The aims of this clinical pilot study are to:

1. to validate the following parameters: mother heart rate, mother ECG, fetal heart rate, contractions, mother oxygen saturation, mother breathing rate, mother blood pressure
2. to evaluate the feasibility on detecting fetal movements
3. to explore how pregnant women and health care professionals perceive the acceptability and usability of the pregnancy monitoring system
4. to explore the possibility to support prenatal attachment between parent and fetus with remote pregnancy monitoring

The participating pregnant women will wear the pregnancy monitoring belt for 2 hours during of which, the data will be collected with pregnancy monitoring belt and patient monitor (reference device). The data from the pregnancy monitoring belt will be compared with the patient monitor data referred as golden standard. The acceptability and usability will be assessed by pregnant women and healthcare professionals by fulfilling a questionnaire and participating in interviews. The data collection will be conducted in hospital environment.

ELIGIBILITY:
Inclusion criteria for pregnant women:

* duration pf pregnancy at least 29+0 weeks
* single pregnancy
* age at least 18 years
* ability to participate in Finnish No exclusion criteria

Inclusion criteria for healthcare professionals:

* being a healthcare professional working with pregnant women
* being able to participate in Finnish No exclusion criteria

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women will be recruited from different units participating in pregnancy care: maternity clinics, pregnancy outpatient clinic and pregnancy follow-up ward. The monitoring during the data collection will not affect the normal pregnancy monitoring practices. The recruitment will be conducted via social media.
  The healthcare professionals will be recruited also from different units in the area of Wellbeing services county of Southwest Finland: pregnancy follow-up ward, labour ward, maternity outpatient clinic and maternity clinics. The recruitment will be conducted via work email.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
fetal heart rate | Two hour data collection
  Fetal heart rate will be measured with the sensorized pregnancy monitoring belt and to evaluate the accuracy of the measurements, the fetal heart rate measurements will be compared with the hospital patient monitor (golden standard).

IPD SHARING:
Plan to Share IPD: Undecided